CLINICAL TRIAL: NCT00003240
Title: A Major Randomised Trial to Determine the Value of Cisplatin-Based Chemotherapy For All Patients With Non-Small Cell Lung Cancer
Brief Title: Standard Therapy Given With or Without Combination Chemotherapy in Treating Patients With Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066115; LLCG-BLT; MRC-BLT; EU-98003
Record Dates: First submitted 1999-11-01; First posted 2004-02-20 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-05

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Ifosfamide; Mitomycin; Vinblastine; Vindesine; Vinorelbine; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: ifosfamide
Drug: mitomycin C
Drug: vinblastine sulfate
Drug: vindesine
Drug: vinorelbine tartrate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not known whether giving chemotherapy in addition to standard therapy is a more effective treatment for lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of standard therapy given with or without combination chemotherapy in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess whether the addition of cisplatin-based chemotherapy to standard treatment improves survival in patients with non-small cell lung cancer.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients undergo primary surgery, radical radiotherapy, radiotherapy with surgery, or best supportive care. Arm II: Patients undergo treatment as in arm I. Beginning within 10 weeks after surgery or radical radiotherapy or as soon as possible after diagnosis, patients receive 1 of the following regimens: Regimen A: Patients receive cisplatin IV on day 1 followed by vindesine on days 1 and 8. Regimen B: Patients receive mitomycin, ifosfamide, and cisplatin on day 1. Regimen C: Patients receive mitomycin, vinblastine, and cisplatin on day 1. Regimen D: Patients receive vinorelbine on days 1 and 8 and cisplatin on day 1. Treatment in all 4 regimens repeats every 3 weeks for 3 courses. Patients are followed at 3 months, 6 months, 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,800 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed non-small cell lung cancer being treated with primary surgery, radical radiotherapy, surgery plus radiotherapy, or best supportive care

PATIENT CHARACTERISTICS: Age: Adult Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: No inadequate renal function Other: No other prior or concurrent malignancy within the past 3 years except nonmelanoma skin cancer Must be fit enough to receive therapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Prior radical radiotherapy allowed Surgery: See Disease Characteristics Prior surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 1995-10

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G. Spiro, Study Chair — University College London Hospitals
Locations (1):
- Middlesex Hospital- Meyerstein Institute, London, England, United Kingdom

REFERENCES:
- [Background] Pignon JP, Tribodet H, Scagliotti GV, et al.: Lung Adjuvant Cisplatin Evaluation (LACE): a pooled analysis of five randomized clinical trials including 4,584 patients. [Abstract] J Clin Oncol 24 (Suppl 18): A-7008, 2006.
- [Result] Brown J, Thorpe H, Napp V, Fairlamb DJ, Gower NH, Milroy R, Parmar MK, Rudd RM, Spiro SG, Stephens RJ, Waller D, West P, Peake MD. Assessment of quality of life in the supportive care setting of the big lung trial in non-small-cell lung cancer. J Clin Oncol. 2005 Oct 20;23(30):7417-27. doi: 10.1200/JCO.2005.09.158. Epub 2005 Sep 12. PMID 16157935
- [Result] Fairlamb DJ, Gower N, Milroy R, et al.: The Big Lung Trial (BLT): determining the value of cisplatin-based chemotherapy for all patients with non-small cell lung cancer (NSCLC). Preliminary results in the radical radiotherapy setting. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2570, 639, 2003.
- [Result] Waller D, Fairlamb DJ, Gower N, et al.: The Big Lung Trial (BLT): determining the value of cisplatin-based chemotherapy for all patients with non-small cell lung cancer (NSCLC). Preliminary results in the surgical setting. [Abstract] Proceedings of the American Society of Clinical Oncology 22 : A-2543, 632, 2003.
- [Result] Stephens RJ, Gower NH, Spiro SG, et al.: The Big Lung Trial (BLT): a major randomised trial to determine the value of cisplatin-based chemotherapy for all patients with non-small cell lung cancer. [Abstract] Lung Cancer 29 (1 Suppl 1): A-61, 20, 2000.